CLINICAL TRIAL: NCT02232204
Title: Sleep in Cardiac Patients With Implantable Cardioverter Defibrillators (ICD)
Brief Title: Sleep and Ventricular Arrhythmias Study
Acronym: SAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 157-2008; R21HL087831 (NIH)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Cardiac Arrhythmia; Implantable Defibrillator User; Insomnia
Keywords: insomnia; implantable cardioverter defibrillator; cardiac arrhythmia; cognitive behavioral treatment
MeSH Terms: conditions — Arrhythmias, Cardiac; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for Insomnia in ICD Patients (CBT-I-ICD) (Active Comparator): Participants will complete 4 weekly therapy sessions focused on improving sleep and reducing ICD-related stress. A multicomponent CBT-I-ICD (Cognitive Behavioral Therapy for Insomnia in ICD Patients) protocol will involve: sleep hygiene, stimulus control, sleep restriction, relaxation, cognitive restructuring, ICD education and recall information, shock planning, and quality of life-improvement recommendations.
  Interventions: Behavioral: CBT for Insomnia in ICD Patients (CBT-I-ICD)
- Waitlist Control (WLC) (No Intervention): Participants in the WLC group will not receive any treatment between the baseline and post-treatment assessments. After the final follow-up assessment, they will be offered the opportunity to receive CBT-I-ICD.

INTERVENTIONS:
Behavioral: CBT for Insomnia in ICD Patients (CBT-I-ICD) — Participants will complete 4 weekly therapy sessions focused on improving sleep and reducing ICD-related stress. A multicomponent CBT-I-ICD (Cognitive Behavioral Therapy for Insomnia in ICD Patients) protocol will involve: sleep hygiene, stimulus control, sleep restriction, relaxation, cognitive restructuring, ICD education and recall information, shock planning, and quality of life-improvement recommendations.
  Arms: CBT for Insomnia in ICD Patients (CBT-I-ICD)

SUMMARY:
This is a single-center, randomized controlled trial study design. Enrolled participants have a cardiovascular condition for which they are undergoing implantable cardioverter defibrillator (ICD) therapy and comorbid insomnia. Participants were randomized to a behavioral intervention for insomnia in ICD patients or a waitlist control. The treatment intervention period lasted 4 weeks with a telephone booster session administered at 3 month follow-up. The objective of the study is to examine the impact of a brief therapy combining established behavioral approaches to treating insomnia with novel components to target negative cognitions and anxieties associated with cardiac disease and ICD implantation. Primary patient outcomes include sleep, psychological functioning, daytime functioning, cardiac functioning, cognitive performance, and ICD adjustment.

DETAILED DESCRIPTION:
Participants will be asked to review the informed consent form and consent to the study prior to beginning any study procedure.

There are six phases of this study: (1) an in-person interview, (2) an in-home single night sleep recording, (3) a two-week baseline period, (4) a 4-week treatment period, (5) a follow-up period immediately after the completion of treatment, (6) and a two-week follow-up period 3-months after the treatment period.

During the interview, participants will be asked questions about their sleep, cardiac, and ICD history. Participants will then visit the University of Florida for a medical history and will be connected to machinery to monitor their sleep. Participants will return home to sleep while still connected to the machine and will return the machine to the University of Florida the next day. A third visit will consist of completing questionnaires and a computerized neurocognitive performance battery to assess several areas of cognitive functioning. Participants will then go home and with brief daily diaries to complete for two weeks while also wearing an actigraph (wristwatch-like device) that measures arm movements to detect sleep/wake during that time.

Participants will then be randomized to (a) the brief cognitive behavioral therapy for insomnia (CBTi) in ICD patients group or (b) the waitlist control group. The treatment consists of 2 weeks of in-person therapy and 2 weeks of therapy conducted over the telephone. Participants assigned to waitlist control will be offered therapy at no cost at the end of the study. Throughout the 4 treatment weeks, participants in both groups will be asked to complete daily sleep diaries.

A follow-up period consisting of two weeks, during which participants will wear the actigraph and complete daily sleep diaries, will take place immediately after treatment completion. Participants will travel to the University two times during this follow-up period in order to pick-up and then return the actigraph and sleep diaries, and will once again complete the questionnaires and neurocognitive testing battery at the end of the 2nd visit. A final follow-up period will occur 3-months following treatment, which will involve visits to the University to pick up the daily sleep diaries and actigraph for sleep monitoring, and then returning these items after completion 2-weeks later. Upon returning the diary and actigraph, participants will complete questionnaires and then be debriefed by study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Current ICD implantation (single or dual lead ICD, ICD and pacemaker)
* Diagnosis of insomnia
* No sleep medications for at least 1 month, or stable on medications for at least 6 months
* Willing to be randomly assigned to treatment
* Able to read and understand English

Exclusion Criteria:

* Sleep disorder other than insomnia
* Significant medical condition other than cardiac disease
* Severe untreated psychopathology
* Neurological disorder
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in subjective and objective sleep | Change from baseline to the two study follow-ups (immediately and 3-months following treatment)
  Sleep diary and actigraphy-derived sleep parameters (averaged over each 14-day data collection period at baseline, post-treatment, and at 3-month follow-up) including: time to fall asleep (sleep onset latency), wake time during the night (waketime after sleep onset), total sleep time, amount of time spent in bed sleeping (sleep efficiency), total nap time, and sleep quality rating.

SECONDARY OUTCOMES:
Change in psychological functioning | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  Changes in reported symptoms of anxiety and depression as assessed by questionnaires from baseline to immediately and 3 months following treatment.
Change in daytime functioning | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  The change in reported insomnia impact, fatigue, and sleepiness as assessed by questionnaires from baseline to immediately and 3 months following treatment.
Change in quality of life | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  The change in reported health-related quality of life as assessed by questionnaires from baseline to immediately and 3 months following treatment.
Change in cardiac functioning | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  The change in device-recorded incidence of ventricular arrhythmia from baseline to immediately and 3 months following treatment.
Change in device adjustment | Change from baseline to the two follow-up periods (immediately and 3-months following treatment
  The change in reported shock anxiety and device-specific acceptance as assessed by questionnaires from baseline to immediately and 3 months following treatment.
Change in cognitive functioning | Change from baseline to immediately after treatment
  The change in computer-recorded cognitive functioning in the domains of executive control, reasoning, working memory, attention, and reaction time as assessed from baseline to immediately following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Aging, Gainesville, Florida, United States